CLINICAL TRIAL: NCT01869309
Title: Overcoming High On-Treatment Platelet Reactivity (HPR) During Prasugrel Therapy
Brief Title: Overcoming High On-Treatment Platelet Reactivity (HPR) During Prasugrel Therapy With Ticagrelor
Acronym: HEIGHTEN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: LifeBridge Health (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2015; ISSBRIL0149 (Other: AstaZeneca)
Record Dates: First submitted 2013-05-28; First posted 2013-06-05 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2013-12

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; anti-platelet medications; Platelet-aggregation Inhibitors
MeSH Terms: conditions — Coronary Artery Disease | interventions — Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-HPR group (No Intervention): The non-HPR group will have PD and genetic testing, with no change in medication.
- HPR Group (Active Comparator): This arm will be split into Group A and Group B which will receive Ticagrelor/Prasugrel in a crossover manner.
  Interventions: Drug: Prasugrel; Drug: Ticagrelor

INTERVENTIONS:
Drug: Prasugrel — Patients will discontinue ticagrelor treatment and start 10 mg prasugrel daily while continuing 81 mg of aspirin daily.
  Arms: HPR Group
Drug: Ticagrelor — Patients will be given 180 mg of Ticagrelor followed by 90 mg twice a day while continuing 81 mg of aspirin daily).
  Arms: HPR Group

SUMMARY:
The primary objective is to determine the pharmacodynamic effect of ticagrelor dosing (180mg LD/ 90mg BID) at 2, 4 hours and 14 days in stable Coronary artery disease (CAD) patients who exhibit high-on prasugrel platelet reactivity defined as Vasodilator Stimulated Phosphoprotein-Phosphorylation (VASP-P) >50%.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female; age ≥ 18 and < 75 years
2. Weight ≥ 60 kg
3. Currently on ASA therapy and eligible to reduce ASA dose to 81 mg daily if on higher dosing
4. On stable prasugrel maintenance dose for ≥1 month
5. Stable CAD patients defined as: subjects with documented evidence of a history of atherosclerotic coronary artery disease/surgical revascularization (defined as either a prior myocardial infarction, percutaneous coronary intervention or coronary artery bypass graft surgery). A minimum of 1 month must have elapsed between a subject's enrolment and any acute event, revascularization procedure or hospitalization for chest pain for that subject.
6. If female, may be enrolled if one of the following 3 criteria are met: 1)Had a hysterectomy or tubal ligation at least 6 months prior to signing ICF, 2)Post-menopausal for at least 1 year, 3)If of childbearing potential, will practice 1 of the following methods of birth control throughout the study: oral, injectable, or implantable hormonal contraceptives; intrauterine device; diaphragm plus spermicide; or female condom plus spermicide. Methods of contraception that are not acceptable are partner's use of condoms or partner's vasectomy.
7. Able and willing to provide written informed consent before entering the study

Exclusion Criteria:

1. Subject plans to undergo coronary revascularization at any time during the trial
2. Presence or history of any of the following: ischemic or hemorrhagic stroke; transient ischemic attack (TIA); intracranial neoplasm; arteriovenous malformation, or aneurysm; intracranial hemorrhage; head trauma (within 3 months of study entry)
3. History of refractory ventricular arrhythmias with an increased risk of bradycardic events (eg, subjects without a pacemaker who have sick sinus syndrome, 2nd or 3rd degree atrioventricular (AV) block or bradycardic-related syncope)
4. History or evidence of congestive heart failure (New York Heart Association Class III or above ≤ 6 months before screening
5. Severe hepatic impairment defined as ALT> 2.5 X ULN
6. Uncontrolled hypertension, or systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg at screening
7. Severely impaired renal function (glomerular filtration rate < 30 mL/minute) or on dialysis
8. Concomitant use with parenteral or oral anticoagulants
9. Platelet count <100 X103

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacodynamic (PD) Vasodilator Stimulated Phosphoprotein-Phosphorylation(VASP-P) in High On Prasugrel Platelet Reactivity(HPPR) stable CAD patients | 2 hours, 4 hours, and 14 days
  The primary objective is to determine the pharmacodynamic effect of ticagrelor dosing (180mg LD/ 90mg BID) at 2, 4 hours and 14 days in stable CAD patients who exhibit high-on prasugrel platelet reactivity defined as VASP-P>50%.

SECONDARY OUTCOMES:
Prevalence of HPPR | 2 hours, 4 hours, and 14 days
  Determine the prevalence of HPPR in a stable PCI population.
CYP2C19 relation to occurence of HPPR | 2 hours, 4 hours, and 14 days
  Determine the relation of CYP2C19 activity to the occurrence of HPPR.
PD VerifyNow in HPPR stable CAD patients | 2 hour, 4 hour, 14 days
  Evaluate the PD effect of ticagrelor dosing (180mg LD/ 90mg BID) at 2, 4 hours and 14 days in stable CAD patients who exhibit HPPR defined as PRU >208 by VerifyNow P2Y12
PD LTA in HPPR stable CAD patients | 2 hours, 4 hours, 14 days
  Evaluate the PD effect of ticagrelor dosing (180mg LD/ 90mg BID) at 2, 4 hours and 14 days in stable CAD patients who exhibit HPPR based on light transmittance aggregometry (5 and 20 uM ADP, 4ug/mL Collagen)
Frequency of HPR | 2 hours, 4 hours, and 14 days
  To determine the frequency of HPR after switching from ticagrelor to prasugrel after 14 days of treatment.
PD effect(Prasugrel) relation to CYP2C19 | 2 hours, 4 hours, and 14 days
  To determine if the PD effect of prasugrel is related to the activity of CYP2C19 (phenotyping and genotyping) by measuring patients with and without HPPR.

OTHER OUTCOMES:
Number of Participants with Adverse Events | 14 days, 28 days
  To evaluate the safety and tolerability of switching subjects from Prasugrel to Ticagrelor and vice versa.

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Gurbel, MD, Principal Investigator — LifeBridge Health
Locations (1):
- Sinai Center for Thrombosis Research, Baltimore, Maryland, United States